CLINICAL TRIAL: NCT05950828
Title: Evaluating the Impact of Online Educator Microskill Training on Educator Knowledge and Skill
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philliber Research & Evaluation (Other)
Responsible Party: Principal Investigator, Ashley Philliber, Managing Director, Philliber Research & Evaluation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Philliberdfusionskillflix
Record Dates: First submitted 2023-07-05; First posted 2023-07-18 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: HIV/AIDS Prevention; STI Prevention; Pregnancy Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SkillTalk (Experimental): Participants will receive one week of access to SkillTalk, a subscription-based microskills video training library designed to enhance the skills of high school sex educators to implement the frequently used core components of sexual and reproductive health (SRH) curricula.
  Interventions: Behavioral: SkillTalk
- Business as usual (No Intervention): Control group will receive "business as usual."

INTERVENTIONS:
Behavioral: SkillTalk — A subscription-based microskills video training library designed to enhance the skills of high school sex educators to implement the frequently used core components of sexual and reproductive health (SRH) curricula.
  Other Names: SkillFlix
  Arms: SkillTalk

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of SkillTalk, a subscription-based microskills video training library designed to enhance the skills of high school sex educators to implement the frequently used core components of sexual and reproductive health (SRH) curricula.

The overall goal of this study is to evaluate the impact of SkillTalk on educators' demonstrable sexual health education skills.

Participants will be asked to:

* Complete a consent form.
* Attend two simulated classroom sessions, either in person or virtually, during which they will teach two prepared lessons that have will be provided to them.
* Be video recorded while teaching.
* Complete a baseline survey and a post-survey.
* If assigned to the treatment group, they will be granted access to SkillTalk for one week to view the videos associated with the answering sensitive questions and using trauma-informed strategies skill sets.

Researchers will compare the treatment group to the control group to see if SkillTalk has an impact on educators' demonstrable sexual health education skills.

ELIGIBILITY:
Inclusion Criteria:

* Teach or have taught groups of youth in a school, clinic or community setting. Group is defined as 4 or more youth. Youth is defined as high school aged youth in grades 9-12.
* Have fewer than three years of experience teaching sexual health education
* Comfortable participating in the role
* Must reside in the U.S.
* Must be at least 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Demonstrable use of microskills | 1 week
  Educators in the intervention group will show greater demonstrable use of microskills than educators in the comparison group. These are rated using a rubric with ratings for each skill from not at all to completely. A total microskills score will be created using this scale of 0 for not at all to 5 for completely. The overall mean score will be the final score with higher scores being more positive outcomes.

SECONDARY OUTCOMES:
Knowledge of microskills | 1 week
  Educators in the intervention group will show greater knowledge of the microskills than educators in the comparison group. A scale will be created based on the SkillTalk site information. An overall percent correct score will be created with higher scores being more positive outcomes.
Self-efficacy and comfort | 1 week
  Educators in the intervention group will show greater self-efficacy and comfort in using microskills than educators in the comparison group. This scale will be created specifically for SkillTalk on a four point scale from strongly disagree to strongly agree with higher scores being more positive outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Philliber Research & Evaluation, Accord, New York, United States

IPD SHARING:
Plan to Share IPD: No